CLINICAL TRIAL: NCT04143906
Title: Randomised, Multicenter Phase II Study in Patients With Metastatic Breast Cancer With Vinorelbine Plus Carboplatin Versus Gemcitabine Plus Carboplatin
Brief Title: Vinorelbine/Carboplatin Versus Gemcitabine/Carboplatin in Metastatic Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Zhiyong Yu, Director of the Breast Surgery, Shandong Cancer Hospital and Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Shandong CHI-10
Record Dates: First submitted 2019-10-27; First posted 2019-10-30 (Actual); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Metastatic Breast Cancer
Keywords: MBC, Vinorelbine, Carboplatin, Gemcitabine, PFS
MeSH Terms: conditions — Breast Neoplasms | interventions — Vinorelbine; Gemcitabine; Carboplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vinorelbine/Carboplatin (Experimental): Vinorelbine 25 mg/m2 d1,8; Carboplatin AUC=6 d1; q 3 weeks
  Interventions: Drug: Vinorelbine; Drug: Carboplatin
- Gemcitabine/Carboplatin (Experimental): Gemcitabine 1000 mg/m2 d1,8; Carboplatin AUC=6 d1; q 3 weeks
  Interventions: Drug: Gemcitabine; Drug: Carboplatin

INTERVENTIONS:
Drug: Vinorelbine — injection
  Arms: Vinorelbine/Carboplatin
Drug: Gemcitabine — injection
  Arms: Gemcitabine/Carboplatin
Drug: Carboplatin — injection

SUMMARY:
Development of an active second-line treatment option for metastatic breast cancer patients previously pre-treated with anthracyclines and taxanes in neoadjuvant, adjuvant or palliative settings. For each randomisation arm, 100 patients will be included. The trial was performed as a 2-stage phase II study according to the optimal design by Simon with overall response rate as the primary objective.

Study Design:

Arm A: Vinorelbine 25 mg/m2 d1,8; Carboplatin AUC=6 d1 q 3 weeks; Arm B: Gemcitabine 1000 mg/m2 d1,8; Carboplatin AUC=6 d1 q 3 weeks;

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed metastatic breast cancer;
2. All patients were required to give written informed consent;
3. To have received a previous treatment with anthracyclines and taxanes;
4. Previous radiotherapy is allowed, whenever the radiated area is not the only disease location;
5. At least 4 weeks since the last previous antineoplastic treatment;
6. Patients must have recovered from all previous toxicities;
7. Karnofsky Performance status >= 70%;
8. Adequate hematological, renal, cardiac and hepatic function;
9. Life expectancy of at least 12 weeks;
10. Patients able to comply and to receive an adequate follow-up;

Exclusion Criteria:

1. Only bone metastases;
2. Active infection;
3. Previous treatment with one of the study drugs;
4. Application of other cytotoxic chemotherapy;
5. Insufficient renal function (creatinine clearance < 60ml/min);
6. Clinically unstable brain metastasis;
7. Pregnancy or lactation;
8. Other primary malignancies (other than carcinoma-in-situ of the cervix or adequately treated basal cell cancer of the skin);
9. Abnormal liver function (bilirubin > 2.0-fold upper normal limit (UNL); Alanine aminotransferase and aspartate aminotransferase >2.5-fold UNL). In patients with hepatic metastasis, a value of Alanine aminotransferase and aspartate aminotransferase of up to 5-fold UNL is permitted;
10. Males;
11. Second malignancy (except for cervix carcinoma in situ or skin carcinoma - no melanoma- with an adequate treatment). Previous malignancies are allowed if disease-free survival is superior to 5 years, except for renal carcinoma or melanoma;

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-10-25 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | Patients enrolled will receive study medication until disease progression, unaccettable toxicity, withdrawal of consent or death, whichever comes first, assested up to 30 months

SECONDARY OUTCOMES:
Overall Survival | Patients enrolled will receive study medication until disease progression, unaccettable toxicity, withdrawal of consent or death, whichever comes first, assested up to 30 months
Clinical Benefit Rate | Patients enrolled will receive study medication until disease progression, unaccettable toxicity, withdrawal of consent or death, whichever comes first, assested up to 30 months
Duration of response | Patients enrolled will receive study medication until disease progression, unaccettable toxicity, withdrawal of consent or death, whichever comes first, assested up to 30 months
Incidence of Treatment-Emergent Adverse Events | Patients enrolled will receive study medication until disease progression, unaccettable toxicity, withdrawal of consent or death, whichever comes first, assested up to 30 months
  Safety of treatment will be evaluated by the frequency of adverse events and serious adverse events, clinically significant abnormal laboratory tests, vital signs, and Eastern Cooperative Oncology Group(ECOG) performance status(PS). All patients who received at least one dose of study treatment will be included in the safety analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Zhiyong Yu, PhD, Study Chair — Shandong Cancer Hospital and Institute; Liang Zhang, MD, Principal Investigator — Shandong Cancer Hospital and Institute